CLINICAL TRIAL: NCT01606761
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study of CNTO 136 (Sirukumab), a Human Anti-IL-6 Monoclonal Antibody, Administered Subcutaneously, in Subjects With Active Rheumatoid Arthritis Despite Anti-TNF-Alpha Therapy
Brief Title: A Study of CNTO 136 (Sirukumab), a Human Anti-IL-6 Monoclonal Antibody, Administered Subcutaneously, in Patients With Active Rheumatoid Arthritis Despite Anti-TNF-Alpha Therapy (SIRROUND-T)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100864; CNTO136ARA3003 (Other: Janssen Research & Development, LLC); 2010-022243-38 (EudraCT Number); U1111-1135-6365 (Other: Universal Trial Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Active rheumatoid arthritis despite anti-TNF-alpha therapy; Sirukumab; Human Anti-IL-6 monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Group 1 (Experimental): Patients will receive placebo every 2 weeks from Week 0 through Week 22, followed by a subcutaneous (SC) sirukumab dose regimen every 2 weeks through Week 52.
  Interventions: Drug: Placebo; Drug: Sirukumab
- Group 2 (Experimental): Patients will receive sirukumab 100 mg SC at Weeks 0, 2, and every 2 weeks through Week 52.
  Interventions: Drug: Sirukumab
- Group 3 (Experimental): Patients will receive sirukumab 50 mg SC at Weeks 0, 4, and every 4 weeks through Week 52. Between sirukumab injections, placebo SC administrations will be made at Weeks 2, 6, and every 4 weeks through Week 52.
  Interventions: Drug: Placebo; Drug: Sirukumab

INTERVENTIONS:
Drug: Placebo — Form=solution for injection, route=subcutaneous use; every 2 weeks from Week 0 through Week 22.
  Arms: Group 1
Drug: Placebo — Form=solution for injection, route=subcutaneous use; Weeks 2, 6, and every 4 weeks through Week 52.
  Arms: Group 3
Drug: Sirukumab — Type=exact, unit=mg, number=50 or 100, form=solution for injection, route=subcutaneous use; every 2 weeks for 100 mg and every 4 weeks for 50 mg, Week 23 through Week 52.
  Arms: Group 1
Drug: Sirukumab — Type=exact, unit=mg, number=100, form=solution for injection, route=subcutaneous use; Weeks 0, 2, and every 2 weeks through Week 52.
  Arms: Group 2
Drug: Sirukumab — Type=exact, unit=mg, number=50, form=solution for injection, route=subcutaneous use; Weeks 0, 4, and every 4 weeks through Week 52.
  Arms: Group 3

SUMMARY:
The purpose of this study is to assess the efficacy of sirukumab as measured by the reduction of the signs and symptoms of rheumatoid arthritis (RA) in patients with active RA who are unresponsive or intolerant to treatment with anti-TNF-alpha agents.

DETAILED DESCRIPTION:
Patients will be randomly assigned to treatment groups, and they and study personnel will not know the identity of the treatments given. Some patients will receive a placebo, which resembles a medication, but does not contain an active substance. This helps to determine if the study agent is effective. Patients will receive placebo or sirukumab by injection under the skin. The expected duration of the study is 68 weeks, which includes 52 weeks of treatment. Participants who complete participation in the study will be eligible for inclusion into the long term extension study if enrollment at a participating site is available to them. If they do not participate in the long-term study, they will continue into the safety follow-up for approximately 16 weeks. The placebo-controlled portion of the study is through Week 24, when placebo patients will cross over to one of two sirukumab dose regimens. Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) for at least 3 months before screening
* Have moderately to severely active RA with at least 4 of 68 tender joints and 4 of 66 swollen joints, at screening and at baseline
* Have had anti-tumor necrosis factor (TNF)-alpha therapy and were unresponsive by 1 of the following 2 reasons: Lack of benefit to at least 1 anti-TNF-alpha biologic therapy, as assessed by the treating physician, after at least 12 weeks of etanercept, yisaipu, adalimumab, golimumab, or certolizumab pegol therapy and/or at least a 14-week dosage regimen (ie, at least 4 doses) of infliximab; Intolerance to at least 2 anti-TNF-alpha biologic therapies, as assessed by the treating physician, to etanercept, yisaipu, adalimumab, golimumab, certolizumab pegol, or infliximab or have documented intolerance to an anti-TNF-alpha agent as described above that precludes further administration of anti-TNF-alpha agents
* If using oral corticosteroids, must be on a stable dose equivalent to less than or equal to 10 mg/day of prednisone for at least 2 weeks prior to the first administration of study agent. If currently not using corticosteroids, must not have received oral corticosteroids for at least 2 weeks prior to the first administration of study agent
* If using non nonsteroidal anti-inflammatory drug (NSAIDs) or other analgesics for RA, must be on a stable dose for at least 2 weeks prior to the first administration of study agent
* If using non-biologic disease modifying antirheumatic drugs (DMARDs) such as methotrexate (MTX), sulfasalazine (SSZ), hydroxychloroquine, chloroquine, or bucillamine, must be on a stable dose for at least 4 weeks prior to the first administration of study agent and should have no serious toxic side effects attributable to the DMARD
* C-reactive protein (CRP) 8.00 mg/L or more or erythrocyte sedimentation rate (ESR) 28 mm/hr or more at screening

Exclusion Criteria:

* Has received infliximab, infliximab biosimilar, or golimumab intravenous (IV) within 8 weeks of the first study agent administration
* Has received subcutaneously (SC) golimumab, adalimumab, or certolizumab pegol within 6 weeks of the first study agent administration
* Has received etanercept or yisaipu within 4 weeks of the first study agent administration
* Has a history of intolerance to tocilizumab that precluded further treatment with it, or inadequate response to 3 months of tocilizumab (anti-IL-6 receptor) therapy. Has used tocilizumab within 8 weeks of the first study agent administration
* Has used B-cell-depleting therapy (eg, rituximab) within 7 months of first study agent administration or have evidence during screening of abnormally low B-cell level caused by previous B-cell depletion therapy
* Has used anakinra within 1 week of first study agent administration
* Has used abatacept or any other biologic therapy for the treatment of RA within 8 weeks of the first study agent administration
* Has received intra-articular (IA), intramuscular (IM), or IV corticosteroids for RA, including adrenocorticotrophic hormone during the 4 weeks prior to first study agent administration
* Has received leflunomide within 24 months before the first study agent administration and has not undergone a drug elimination procedure, unless the M1 metabolite is measured and is undetectable
* Has a history of cyclophosphamide or cytotoxic agent use
* Has received cyclosporine A, azathioprine, tacrolimus, mycophenolate mofetil, oral or parenteral gold, or D-penicillamine within 4 weeks of the first study agent administration
* Has received an investigational drug (including investigational vaccines) or used an investigational medical device within 3 months or 5 half-lives, whichever is longer, before the first study agent administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2016-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (201):
- United States (81):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Covina, California
  - El Cajon, California
  - Hemet, California
  - Huntington Beach, California
  - La Jolla, California
  - La Palma, California
  - Placentia, California
  - Santa Monica, California
  - Tustin, California
  - Upland, California
  - Victorville, California
  - Whittier, California
  - Hamden, Connecticut
  - Aventura, Florida
  - Boca Raton, Florida
  - Brandon, Florida
  - Daytona Beach, Florida
  - Lake Mary, Florida
  - Miami, Florida
  - Naples, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Bowling Green, Kentucky
  - Monroe, Louisiana
  - Shreveport, Louisiana
  - Cumberland, Maryland
  - Frederick, Maryland
  - Hagerstown, Maryland
  - Eagan, Minnesota
  - Rochester, Minnesota
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Freehold, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Lake Success, New York
  - Plainview, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Edmond, Oklahoma
  - Tulsa, Oklahoma
  - Erie, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wyomissing, Pennsylvania
  - East Greenwich, Rhode Island
  - Charleston, South Carolina
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Cypress, Texas
  - Dallas, Texas
  - Houston, Texas
  - Katy, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Richmond, Texas
  - Victoria, Texas
  - Kennewick, Washington
  - Seattle, Washington
  - Beckley, West Virginia
  - Clarksburg, West Virginia
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Miguel de Tucumán
- Australia (2):
  - Campbelltown
  - Victoria Park
- Vienna, Austria
- Liège, Belgium
- Canada (7):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Kitchener, Ontario
  - Burlington
  - St. John's
  - Toronto
- Zagreb, Croatia
- France (2):
  - Paris
  - Toulouse
- Germany (13):
  - Berlin
  - Cologne
  - Dresden
  - Erfurt
  - Frankfurt am Main
  - Gÿttingen N/A
  - Hamburg
  - Herne
  - Kiel Kronshagen
  - Schwerin
  - Vogelsang-Gommern
  - Würzburg
  - Zerbst
- Japan (39):
  - Ayauta
  - Bunkyō City
  - Fukuoka
  - Fukuyama
  - Higashihiroshima
  - Hiroshima
  - Izumo
  - Kagoshima
  - Katō
  - Kawagoe
  - Kita-Gun
  - Kumamoto
  - Kurume
  - Matsuyama
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nagoya
  - Nishimuro-Gun
  - Nishinomiya
  - Okayama
  - Osaka
  - Sapporo
  - Sasebo
  - Shibata
  - Shimonoseki
  - Shimotsuke
  - Shinjuku-Ku
  - Sumida-Ku
  - Takaoka,Toyama
  - Takasaki
  - Tokorozawa
  - Tokushima
  - Tomakomai
  - Tomishiro
  - Tonami
  - Tsu
  - Ureshino
  - Yokohama
- Lithuania (2):
  - Kaunas
  - Klaipėda
- Mexico (3):
  - Guadalajara
  - Mérida
  - San Luis Potosí City
- Sneek, Netherlands
- New Zealand (3):
  - Christchurch
  - Hamilton
  - Wellington
- Poland (6):
  - Bydgoszcz
  - Elblag
  - Lublin
  - Poznan
  - Ustroń
  - Warsaw
- Portugal (2):
  - Coimbra
  - Lisbon
- San Juan, Puerto Rico
- Russia (9):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Omsk
  - Orenburg
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Ulyanovsk
- South Korea (9):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Seongnam-si
  - Seoul
  - Suwon
- Spain (7):
  - A Coruña
  - Bilbao
  - Madrid
  - Mérida
  - San Cristóbal de La Laguna
  - Santander
  - Santiago de Compostela
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (5):
  - Barnsley
  - London
  - Middlesbrough
  - Sheffield
  - Wigan

REFERENCES:
- [Derived] Aletaha D, Bingham CO 3rd, Tanaka Y, Agarwal P, Kurrasch R, Tak PP, Popik S. Efficacy and safety of sirukumab in patients with active rheumatoid arthritis refractory to anti-TNF therapy (SIRROUND-T): a randomised, double-blind, placebo-controlled, parallel-group, multinational, phase 3 study. Lancet. 2017 Mar 25;389(10075):1206-1217. doi: 10.1016/S0140-6736(17)30401-4. Epub 2017 Feb 16. PMID 28215362

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 878 participants (placebo [n=294], sirukumab 50 mg every 4 week (q4w) [n=292], and sirukumab 100 milligram (mg) every 2 week (q2w) [n=292]) were randomized and included in the study.
Groups:
- Placebo: Participants received matching placebo every 2 week (q2w) until either early escape (EE) at Week 18, or crossed over (CO) at Week 24. Participants who met EE criteria at Week 18 or crossover (CO) at Week 24 re-randomized and received subcutaneous (SC) sirukumab 50 mg dose regimen q4w up to Week 52. Participants who discontinued or completed study agent administration before and up to Week 52 entered the safety follow-up period as well as those who completed through Week 52 were followed up for safety.
- Sirukumab 50 mg q4w: All participants received Sirukumab 50 mg SC at Week 0, 4 and q4w up to Week 52. Participants who discontinued or completed study agent administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- Sirukumab 100 mg q2w: All participants received Sirukumab 100 mg SC at Week 0, 2 and q2w up to Week 24. Participants who received matching placebo in the placebo controlled period and met EE criteria at Week 18 or crossover (CO) at Week 24 re-randomized and received subcutaneous (SC) sirukumab 100 mg dose regimen q2w up to Week 52. Participants who discontinued or completed study agent administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- Placebo to 50 mg q4w Due to EE or CO: Participants who received matching placebo in the placebo controlled period were re-randomized (due to early escape [EE] at Week 18 or crossed over [CO] at Week 24) to receive subcutaneous (SC) sirukumab 50 mg dose regimen q4w up to Week 52. Participants who discontinued or completed study agent administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- Placebo to 100 mg q2w Due to EE or CO: Participants who received matching placebo in the placebo controlled period were re-randomized (due to EE at Week 18 or CO at Week 24) to receive subcutaneous (SC) sirukumab 100 mg dose regimen q2w up to Week 52. Participants who discontinued or completed study agent administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
Period: Prior to Week 24
Arm/Group | Placebo | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Placebo to 50 mg q4w Due to EE or CO | Placebo to 100 mg q2w Due to EE or CO
Started | 294 | 292 | 292 | 0 | 0
Participants Re-randomized at Week 18 | 94 (Out of 94, 46 were re-randomized to sirukumab 50 mg and 48 were re-randomized to 100 mg group.) | 0 | 0 | 0 | 0
Completed | 252 | 237 | 245 | 0 | 0
Not Completed | 42 | 55 | 47 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 10 | 9 | 0 | 0
Not completed — Adverse Event | 11 | 18 | 22 | 0 | 0
Not completed — Lack of Efficacy | 15 | 14 | 8 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 1 | 0 | 0
Not completed — Other | 4 | 7 | 5 | 0 | 0
Period: Week 24 to Week 52
Arm/Group | Placebo | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Placebo to 50 mg q4w Due to EE or CO | Placebo to 100 mg q2w Due to EE or CO
Started | 0 | 237 | 245 | 126 (Participants re-randomized at Week 18 (46) and Week 24 (80) were included.) | 126 (Participants re-randomized at Week 18 (48) and Week 24 (78) were included.)
Treated | 0 | 237 | 245 | 124 | 126
Completed | 0 | 204 | 212 | 109 | 106
Not Completed | 0 | 33 | 33 | 17 | 20
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 11 | 14 | 3 | 15
Not completed — Death | 0 | 0 | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 13 | 7 | 10 | 3
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 5 | 2 | 2
Period: Safety Follow-up Period (Week 52-68)
Arm/Group | Placebo | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Placebo to 50 mg q4w Due to EE or CO | Placebo to 100 mg q2w Due to EE or CO
Started | 28 | 65 | 62 | 9 | 19
Safety Population | 28 | 65 | 62 | 7 | 19
Completed | 24 | 55 | 45 | 7 | 11
Not Completed | 4 | 10 | 17 | 2 | 8
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 6 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 3 | 9 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Total
Number analyzed (Participants) | 294 | 292 | 292 | 878
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (12.19) | 0 (11.89) | 0 (12.28) | 0
  Between 18 and 65 years | 228 | 225 | 230 | 683
  >=65 years | 66 | 67 | 62 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.19) | 55.8 (11.89) | 55 (12.28) | 55.4 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 232 | 240 | 712
  Male | 54 | 60 | 52 | 166
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 10 | 6 | 3 | 19
  Australia | 1 | 2 | 0 | 3
  Austria | 2 | 0 | 0 | 2
  Belgium | 1 | 0 | 0 | 1
  Canada | 2 | 7 | 1 | 10
  France | 0 | 1 | 0 | 1
  Germany | 7 | 13 | 7 | 27
  Italy | 5 | 0 | 4 | 9
  Japan | 37 | 35 | 44 | 116
  Lithuania | 4 | 7 | 5 | 16
  Mexico | 7 | 4 | 6 | 17
  Netherlands | 4 | 1 | 1 | 6
  Poland | 21 | 29 | 26 | 76
  Portugal | 3 | 4 | 4 | 11
  Puerto Rico | 1 | 6 | 1 | 8
  Republic of Korea | 5 | 7 | 5 | 17
  Russian Federation | 18 | 11 | 21 | 50
  Spain | 8 | 8 | 7 | 23
  Taiwan, Province of China | 8 | 2 | 2 | 12
  United Kingdom | 2 | 4 | 3 | 9
  United States | 148 | 145 | 152 | 445

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Response at Week 16
Description: The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 scale, 0 =no pain and 10 =worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 =no pain to 10 =worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Week 16
Population: Efficacy full analysis set included all participants who were randomized into the study.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received matching placebo every 2 week (q2w) until either early escape (EE) at Week 18, or crossed over (CO) at Week 24. Participants who met EE criteria at Week 18 or crossover (CO) at Week 24 re-randomized and received subcutaneous (SC) sirukumab 50 mg dose regimen q4w up to Week 52.
- Sirukumab 50 mg: Participants received Sirukumab 50 mg SC at Week 0, 4 and q4w up to Week 52.
- Sirukumab 100 mg: Participants received Sirukumab 100 mg SC at Week 0, 2 and q2w up to Week 24. Participants who received matching placebo in the placebo controlled period and met EE criteria at Week 18 or crossover (CO) at Week 24 re-randomized and received subcutaneous (SC) sirukumab 100 mg dose regimen q2w up to Week 52.
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 294 | 292 | 292
Percentage of Participants | 24.1 | 40.1 | 45.2
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 15.9, 95% CI 2-sided [8.5 to 23.2]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 21.0, 95% CI 2-sided [13.6 to 28.5]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Week 24
Population: Efficacy full analysis set included all participants who were randomized into the study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 294 | 291 | 292
Units on a scale
  Baseline | 1.5663 (0.65223) | 1.6499 (0.59743) | 1.6122 (0.61320)
  Change at Week 24 | -0.12 (0.491) | -0.31 (0.543) | -0.33 (0.526)
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Square (LS) mean difference = -0.17, 95% CI 2-sided [-0.251 to -0.088]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.194, 95% CI 2-sided [-0.275 to -0.112]

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 50 Response at Week 24
Description: The ACR 50 Response is defined as >= 50 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS ( 0-10 scale, 0 =no pain and 10 =worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 =no pain to 10 =worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Efficacy full analysis set included all participants who were randomized into the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 294 | 292 | 292
Percentage of Participants | 8.8 | 20.9 | 21.6
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 12.0, 95% CI 2-sided [6.4 to 17.7]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 12.7, 95% CI 2-sided [7.0 to 18.4]

4. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (CRP) Remission at Week 24
Description: The Disease Activity Index Score 28 (DAS28) based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS28 (CRP) remission is defined as a DAS28 (CRP) value of less than (<) 2.6 at any study visit.
Time Frame: Week 24
Population: Efficacy full analysis set included all participants who were randomized into the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 294 | 292 | 292
Percentage of Participants | 8.2 | 19.2 | 21.6
Statistical Analysis 1: Comparison: Placebo vs Sirukumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 11.0, 95% CI 2-sided [5.5 to 16.5]
Statistical Analysis 2: Comparison: Placebo vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 13.4, 95% CI 2-sided [7.8 to 19.1]

ADVERSE EVENTS:
Time Frame: Up to Week 68
Description: For treatment period (up to Week 52), safety population (SP) included all participants who received at least 1 partial or complete dose of study agent. For safety follow-up (SFU) (Week 52-68), SP included participants who decided to enter in safety follow-up period and had at least 1 SFU visit after the discontinuation of study agent (Week 52-68).
Groups:
- Week (W) 24-Placebo: Participants received matching placebo every 2 week (q2w) until either early escape (EE) at Week 18, or crossover (CO) at Week 24.
- W24 to W52-Placebo to 50 mg q4w Due to EE or CO: Participants who received matching placebo in the placebo controlled period and were re-randomized (due to early escape [EE] at Week 18 or crossed over [CO] at Week 24) to receive subcutaneous (SC) sirukumab 50 mg q4w dose regimen up to Week 52.
- W52-Sirukumab 50 mg q4w: Participants received Sirukumab 50 mg SC at Week 0, 4 and q4w up to Week 52.
- W24 to W52-Placebo to 100 mg q2w Due to EE or CO: Participants who received matching placebo in the placebo controlled period and were re-randomized (due to early escape [EE] at Week 18 or crossed over [CO] at Week 24) to receive subcutaneous (SC) sirukumab 100 mg q4w dose regimen up to Week 52.
- W52-Sirukumab 100 mg q2w: Participants received sirukumab 100 mg SC at Week 0, 2 and q2w up to Week 52.
- W52 to W68-Placebo: Participants who discontinued or completed study agent administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- W52 to W68-Placebo to 50 mg q4w Due to EE or CO: Participants who discontinued or completed sirukumab 50 mg q4w due to EE or CO administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- W52 to W68-Sirukumab 50 mg q4w: Participants who discontinued or completed sirukumab 50 mg q4w administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- W52 to W68-Placebo to 100 mg q2w Due to EE or CO: Participants who discontinued or completed sirukumab 100 mg q2w due to EE or CO administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
- W52 to W68-Sirukumab 100 mg q2w: Participants who discontinued or completed sirukumab 100 mg q2w administration up to Week 52 and decided to enter the safety follow-up period were followed up for safety from Week 52 to Week 68.
Arm/Group | Week (W) 24-Placebo | W24 to W52-Placebo to 50 mg q4w Due to EE or CO | W52-Sirukumab 50 mg q4w | W24 to W52-Placebo to 100 mg q2w Due to EE or CO | W52-Sirukumab 100 mg q2w | W52 to W68-Placebo | W52 to W68-Placebo to 50 mg q4w Due to EE or CO | W52 to W68-Sirukumab 50 mg q4w | W52 to W68-Placebo to 100 mg q2w Due to EE or CO | W52 to W68-Sirukumab 100 mg q2w
Serious Adverse Events (participants affected / at risk) | 15/294 | 8/124 | 51/292 | 18/126 | 37/292 | 0/28 | 0/7 | 1/65 | 2/19 | 0/62
Other Adverse Events (participants affected / at risk) | 106/294 | 50/124 | 152/292 | 63/126 | 169/292 | 0/28 | 1/7 | 2/65 | 3/19 | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week (W) 24-Placebo (N=294) | W24 to W52-Placebo to 50 mg q4w Due to EE or CO (N=124) | W52-Sirukumab 50 mg q4w (N=292) | W24 to W52-Placebo to 100 mg q2w Due to EE or CO (N=126) | W52-Sirukumab 100 mg q2w (N=292) | W52 to W68-Placebo (N=28) | W52 to W68-Placebo to 50 mg q4w Due to EE or CO (N=7) | W52 to W68-Sirukumab 50 mg q4w (N=65) | W52 to W68-Placebo to 100 mg q2w Due to EE or CO (N=19) | W52 to W68-Sirukumab 100 mg q2w (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecal Incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Pseudocyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Device Dislocation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impaired Healing (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Jaw (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis Infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 5 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection Pseudomonas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Morganella Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intermittent Claudication (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosed Varicose Vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week (W) 24-Placebo (N=294) | W24 to W52-Placebo to 50 mg q4w Due to EE or CO (N=124) | W52-Sirukumab 50 mg q4w (N=292) | W24 to W52-Placebo to 100 mg q2w Due to EE or CO (N=126) | W52-Sirukumab 100 mg q2w (N=292) | W52 to W68-Placebo (N=28) | W52 to W68-Placebo to 50 mg q4w Due to EE or CO (N=7) | W52 to W68-Sirukumab 50 mg q4w (N=65) | W52 to W68-Placebo to 100 mg q2w Due to EE or CO (N=19) | W52 to W68-Sirukumab 100 mg q2w (N=62)
Blepharitis (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 10 | 1 | 13 | 0 | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 4 | 5 | 28 | 19 | 47 | 0 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 2 | 4 | 8 | 10 | 31 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 2 | 4 | 7 | 24 | 0 | 0 | 0 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 7 | 13 | 4 | 22 | 0 | 1 | 0 | 0 | 0
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 2 | 34 | 7 | 26 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 2 | 5 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 8 | 5 | 14 | 3 | 15 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 6 | 24 | 9 | 26 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 11 | 2 | 13 | 6 | 19 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 6 | 12 | 27 | 8 | 23 | 0 | 0 | 1 | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 4 | 6 | 18 | 5 | 15 | 0 | 0 | 1 | 1 | 1
Hepatitis B Dna Assay Positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil Count Increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
X-Ray with Contrast Upper Gastrointestinal Tract Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 1 | 9 | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5 | 1 | 7 | 0 | 1 | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 28 | 13 | 30 | 4 | 30 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 13 | 4 | 22 | 0 | 1 | 0 | 0 | 0
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 9 | 0 | 15 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 7 | 3 | 17 | 3 | 15 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.